CLINICAL TRIAL: NCT05574686
Title: Tracking Social Outcomes of Hypertension in Women With Breast Cancer
Brief Title: Telemonitoring Hypertension and Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Cheryl Clark, MD, ScD (Unknown); Saurabh Chandra, MD (Unknown); Richard Summers, MD (Unknown)
Responsible Party: Principal Investigator, LaQuita Cooper, PhD, MPH, MHSA, Program Manager, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMMCHTNBC
Record Dates: First submitted 2022-10-04; First posted 2022-10-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Breast Cancer
MeSH Terms: conditions — Hypertension; Breast Neoplasms | interventions — Food Insecurity

STUDY DESIGN:
Intervention Model Description: Using the telemonitoring kit of iPad to access daily health sessions and remote blood pressure cuff to monitor blood pressure measurements. Patients will then obtain a BP measurement using the appropriate technique described above. Patients are asked to obtain two consecutive BP measurements during each session and register at least 6 sessions per week. Every 2 weeks, BP measurements will be assessed.
Masking Description: No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telehealth Hypertension and Food Insecurity Intervention (Experimental): Telehealth Hypertension and Food Insecurity Intervention Established clinical telehealth services will be provided to monitor and give behavioral and educational management advice to women with breast cancer to better control their hypertension. Resources for food insecurity will be provided to participants.
  Interventions: Behavioral: Telehealth Blood Pressure Monitoring and Food Insecurity

INTERVENTIONS:
Behavioral: Telehealth Blood Pressure Monitoring and Food Insecurity — Telehealth Blood Pressure Monitoring and Food Insecurity

SUMMARY:
The goal of this clinical trial-prospective study will provide important information on equitable implementation strategies to improve hypertension management in women with breast cancer by evaluating the feasibility and safety of remote hypertension management using home blood pressure telemonitoring that will provide individualized hypertension management, health and wellness education for hypertension prevention of women with breast cancer stages I-IV. Also this study may provide evidence to inform a potential paradigm shift in joint social and clinical management of hypertension that future studies may use to address complex social and clinical comorbidities that affect women with hypertension in Mississippi. The main questions this study aims to answer are:

1. To examine the feasibility of using home BP telemonitoring to provide individualized hypertension management in a population of women with breast cancer and food insecurity.
2. To examine the effectiveness of telemonitoring in achieving 2017 ACC/AHA guidelines for hypertension control in women with breast cancer and food insecurity using the RE-AIM framework.
3. To pilot the integration of a community service partnership to decrease food insecurity in the 40 women who participate in the home BP telemonitoring program.

Using the mailed telemonitoring kit (iPad tablet and Blood Pressure Cuff) the participants of this study will be asked to access a daily health session using iPad and obtain a blood pressure measurement using blood pressure cuff that transmits readings wirelessly via Bluetooth to the tablet which is uploaded directly to the participants UMMC electronic health records. Participants are asked to obtain two consecutive blood pressure measurements during each session and register at least 6 sessions per week. The study duration will be 6 months. Every 2 weeks blood pressure measurements will be assessed. If less than 75% of measurements are at goal systolic blood pressure 75% of measurements are at goal systolic blood pressure<130mmHg and diastolic blood pressure <80mmHg, the patients nurse coordinator will contact them via telephone and assess for medication adherence and report to the patient's primary care provider and oncologist.

DETAILED DESCRIPTION:
This is a prospective pilot study with collaborating sites of UMMC Cancer Center Research Institute, UMMC Cancer Treatment Center, UMMC Center for National Telehealth Center for Excellence and UMMC Myrlie Evers-Williams Institute for the Elimination of Health Disparities. The study aims to evaluate the feasibility and safety of remote hypertension management using a home blood pressure telemonitoring to provide individualized hypertension management, health and wellness education for hypertension prevention of women with breast cancer stages I-IV in Mississippi at the UMMC Cancer Treatment Center. Additionally, the study will examine the effectiveness of remote hypertension management using home BP telemonitoring in achieving BP control with 2017 ACC/AHA guidelines. Further, the study will assess the social determinant of health screening and service connection with UMMC EversCare and is a part of Myrlie Evers-Williams Institute for Elimination of Health Disparities to decrease food insecurity in 40 women patients who participate in the remote hypertension management monitoring pilot project using home BP telemonitoring program.

Patients with breast cancer and elevated BP, as identified by UMMC electronic health record, will be initially recruited for study enrollment and obtain informed consent by Breast Oncologist and/or Primary Care Providers. The patients will then be contacted by Telehealth Nurse Coordinator and/or Research Specialist via telephone to confirm consent of participation, awareness of who will be their contact through-out the study and confirm address to mail telemonitoring kit. Patients will be mailed a telemonitoring kit including an iPad tablet equipped with a wireless BP cuff that transmits measurements directly to the UMMC EHR and monitored by the UMMC Center for Telehealth. Consenting patients will participate in a 6-month intervention period during which they will transmit daily blood pressure recordings with regular contact by a Telehealth Nurse Coordinator who will also provide education and encourage healthy lifestyle habits. Study patients will be instructed to access a daily "health session" which begins by asking two questions include: 1) "Have you taken your medications in the past 24 hours?" and 2) "Are you having any problems that you would like your nurse coordinator to call you about before the next scheduled call?" Patients will then obtain a BP measurement using the appropriate technique. Patients are asked to obtain two consecutive BP measurements during each session and register at least 6 sessions per week. Patients are encouraged to equally divide daily health sessions between the morning and evenings and patients may register more than one session per day. If less than 75% of measurements are at goal systolic BP <140 mmHg and diastolic BP <90 mmHg, the patient's Telehealth Nurse Coordinator will contact them and assess for medication adherence and report to the patients Breast Oncologist and/or Primary Care Provider.

The Breast Oncologist and/or Primary Care Provider will be provided with a monthly report of the patient's progress including medication, biometric information and any hospital or clinic visits. Food resource provision. Implementation procedures for providing food resources will be tailored and evaluated in partnership with UMMC Ambulatory EversCare-MEWI. Data analysis will track metrics of study enrollment, study completion, safety and BP change from baseline. Much of the study protocol is based on a recently published clinical trial demonstrating significantly improved BP control using home BP telemonitoring as compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility and exclusion criteria are intended to capture a population broadly representative of breast cancer patient's stages I-IV with hypertension, while excluding patients with hypertension complicated by major co-morbidities as determined by chart review who would not be appropriate for algorithmic management.
* Clinical/study eligibility will be confirmed by the patient's Breast Oncologist and/or Primary Care Providers who will refer identified patients or provide permission for outreach to eligible patients for recruitment into the pilot study.
* Patients eligible for the intervention must meet all eligibility criteria intended to identify breast cancer patients with hypertension and positive screening for food insecurity according to the 2017 ACC/AHA Guidelines, healthcare provider hypertension diagnosis and Hunger Vital Signs Tool United States Departments of Agriculture:
* Women ages 18 years and older UMMC breast cancer patients in stages I-IV as primary diagnosis within the last three years and who were diagnosed with hypertension exceeding 2017 ACC/AHA guidelines of ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg will be identified from UMMC electronic health records (EHR).
* Women ages 18 years and older UMMC breast cancer patients in stages I-IV as a primary diagnosis within the last three years with physician-coded hypertension, who have their most recently documented blood pressures exceeding 2017 ACC/AHA guidelines of ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg in at least three consecutive instances in the EHR, three consecutive high BP measurements within 12 months, consistent with SNOMED coded phenotypes for hypertension identify from UMMC EHR records (A diagnosis of hypertension).
* Positive screening for food insecurity via the Hunger Vital Signs tool, a validated two-question screening tool based on the United States Department of Agriculture.
* Ability to speak English.
* Reliable access to internet, video and telephone services.

Exclusion Criteria:

* Stage 4 or 5 kidney disease (eGFR <30 ml/min/1.73m2 on the most recent measurement)
* Acute coronary syndrome, coronary revascularization, stroke, or other major cardiovascular event within the past 3 months
* Known secondary causes of hypertension including coarctation of the aorta, pheochromocytoma, and adrenal cortical hypertension
* Prescribed 3 or more antihypertensive medications
* Class III or IV New York Heart Association heart failure or left ventricular ejection fraction <50%
* Institutionalized (i.e., nursing home) or limited life expectancy as determined by chart review including advanced stage cancer, severe frailty, or other major comorbidity
* Further exclusion criteria include unwillingness to be followed for the duration of the study, participation in another clinical trial or research study, difficulty with communication in English without an interpreter over the telephone, substance abuse, dementia, disability or mental illness that would prohibit ability to provide informed consent or perform home BP monitoring. Additionally, patients are ineligible if they report a major health event requiring hospitalization since the last documented UMMC clinic visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females sex assigned at birth
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Control | 6-months
  The study will provide new and important insights into remote hypertension management using telehealth monitoring from a remote blood pressure cuff. This represents a potential paradigm shift in the ability to move effectively manage hyperextension and other chronic disease on a large scale. The study aims to reduce blood pressure through a comprehensive remote hypertension management program. Participants stand to gain significant benefit from hypertension control. this program is intended to control hypertension without any additionally scheduled clinic visits, and therefore study patients stand to realize the benefit of time and opportunity costs not spent traveling and attending clinic visits.

SECONDARY OUTCOMES:
Decrease Food Insecurity | 6 months
  Decreasing food insecurity through social resource connections. Implementation procedures for providing healthy food resources will be tailored and evaluated. The participants will participate in a health education session via iPad that includes blood pressure management and healthy eating. The participants will be provided with resources to receive healthy foods as an approach to lifestyle change of diet to decrease complications of stroke, heart failure, heart attack and kidney damage. Making dietary changes are effective treatments for reducing high blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mississippi Medical Center Cancer Institute, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
individual data will only be shared with investigators on the current study.

REFERENCES:
- [Background] Mendy VL, Rowell-Cunsolo T, Bellerose M, Vargas R, Zhang L, Enkhmaa B. Temporal Trends in Hypertension Death Rate in Mississippi, 2000-2018. Am J Hypertens. 2021 Sep 22;34(9):956-962. doi: 10.1093/ajh/hpab068. PMID 33954415
- [Background] Berkowitz SA, Basu S, Gundersen C, Seligman HK. State-Level and County-Level Estimates of Health Care Costs Associated with Food Insecurity. Prev Chronic Dis. 2019 Jul 11;16:E90. doi: 10.5888/pcd16.180549. PMID 31298210
- [Background] Williams MS, Beech BM, Griffith DM, Jr Thorpe RJ. The Association between Hypertension and Race/Ethnicity among Breast Cancer Survivors. J Racial Ethn Health Disparities. 2020 Dec;7(6):1172-1177. doi: 10.1007/s40615-020-00741-7. Epub 2020 Mar 17. PMID 32185742